CLINICAL TRIAL: NCT05239442
Title: Engaging Elderly People Living in Institutions in Eating Situations
Acronym: ENGAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VAN WYMELBEKE I-SITE 2017
Record Dates: First submitted 2021-10-27; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Under-consumption of Food

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients (Other): Hospital Patients:
  - Person hospitalized in one of the following departments: endocrinology-diabetology, geriatric medicine, pulmonology, rheumatology, dermatology, infectious diseases, internal medicine, cardiology, as well as in the rehabilitation department
  Interventions: Other: Taste Commission; Other: Evaluation of the taste commissions
- Institutional staff (Other): Person working in the establishment where the taste commissions have been in place for at least 3 months
  Interventions: Other: Entretien SWOT
- Residents (Other): Patients residing in nursing home
  Interventions: Other: Taste Commission; Other: Evaluation of the taste commissions; Other: Entretien SWOT

INTERVENTIONS:
Other: Taste Commission — Evaluation of the daily meal once a week:
  Introduction on the different sensory dimensions of the food, hedonic rating for each component, indicate what pleases/what could be improved in the recipe.
  Arms: Patients; Residents
Other: Evaluation of the taste commissions — At 0, 3, 6 months:
  * Food intake measurement, satisfaction measurement, and food waste measurement performed on 2 days (same week but not necessarily consecutive)
  * Assessment of nutritional status using the Mini-Nutritional Assessment (MNA)
  Arms: Patients; Residents
Other: Entretien SWOT — Individual semi-guided face-to-face interview with an experimenter. They will allow us to identify the positive and negative effects of the taste commissions in the establishment as well as the levers and difficulties encountered during the implementation of the taste commissions. These interviews will be recorded using an audio device (dictaphone). Their content will then be transcribed in full.
  Arms: Institutional staff; Residents

SUMMARY:
Several recent studies have revealed a significant under-consumption of food in hospitals and nursing homes. For instance, at the Dijon University Hospital, 8 out of 10 patients consume less than 80% of the meals served. This has two consequences: an increase in the risk of malnutrition (some patients leave the hospital in such a poor nutritional state that they must be re-hospitalized within six months) and significant food waste. At the heart of this problem, the taste of the food is the subject of frequent and recurrent complaints from users. Although the food industry widely uses sensory methods to adapt its products to the taste of consumers, these methods are rarely used by the organizations that provide meals to care institutions.

The objective is to establish "taste commissions" in the daily practice in institutions for the elderly (hospital, nursing home), in order to improve the organoleptic quality of the meals served according to the expectations and preferences of the users. The principle of this system is to allow the users to taste the dishes produced by the kitchen of the establishment and to transmit these evaluations to the cooks so that they can rework the recipes according to the users' feedback.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized patients:

* Person hospitalized in one of the following departments: the endocrinology-diabetology department, geriatric medicine, pulmonology, rheumatology, dermatology, infectious diseases, internal medicine, cardiology, as well as the rehabilitation department, which are departments with an average length of stay sufficient to perform the study
* Person aged ≥ 50 years (this choice was made because more than 60% of the hospitalized population is currently over 50 years old)
* Person having given their oral agreement
* Person with an oral diet and eating without assistance
* Person with a normal texture diet
* For taste commissions and SWOT interviews: person with sufficient cognitive status to answer questions in a questionnaire or interview (MMSE > 21).

Residents in nursing home (EHPAD):

* Person residing in EHPAD
* Person aged ≥ 65 years
* Person having given oral consent
* Person who is orally fed and self-feeding
* Person with a normal texture diet
* For taste commissions and SWOT interviews: person with sufficient cognitive status to answer questions in a questionnaire or interview (MMSE > 21).

Facility staff for SWOT interviews:

* Person who has worked at the facility where the taste commissions were implemented at least 3 months previously.
* Person who gave oral consent
* Person between the ages of 18 and 60

Exclusion Criteria:

* Person at the end of life
* Person with an eating disorder
* Person with a significant chronic psychiatric disorder (psychosis, manic-depression).
* Person requiring enteral or parenteral nutrition.
* Person in a period of exclusion from a previous study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
weight of consumed ingesta | Change from Baseline to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France